CLINICAL TRIAL: NCT04810845
Title: Clinical Use of the SmartCardia Wireless Recorder for the Detection of Myocardial Ischemia in the Setting of Coronary Artery Disease: a Single Arm, Prospective Trial
Brief Title: SmartCardia for the Detection of Myocardial Ischemia in Coronary Artery Disease
Acronym: Smartschemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Niccolo' Maurizi, MD, Cardiology Fellow, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-0000
Record Dates: First submitted 2021-02-21; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Myocardial Ischemia
Keywords: ischemia
MeSH Terms: conditions — Myocardial Ischemia; Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing coronary angiography with planned PCI (Experimental): Patients with a known coronary artery disease admitted for elective coronary angiography with planned PCI would be enrolled
  Interventions: Device: Application of Class II A device SmartCardia

INTERVENTIONS:
Device: Application of Class II A device SmartCardia — Application of SmartCardia monitor patch 30 minutes before coronary angiography (2/3 devices per-patients would be applied). Non invasive recording of single-lead ECG, respiratory rate, pulse transit time, heart rate would occur pre, during and post (30 minutes) primary angioplasty procedure
  Other Names: SmartCardia multiparametric Device

SUMMARY:
Coronary artery disease and myocardial ischemia are among the leading causes of death and disability in the Westerns countries. Timely and accurate diagnosis of myocardial ischemia at the moment of symptom onset is crucial and often delayed. Portable smart medical devices nowadays offers the possibility of ubiquitous self multi-parametric monitoring. Application of such technologies to timely and autonomous detection of myocardial ischemia could be an effective strategy to an earlier and better treatment of symptomatic coronary artery disease.

The primary objective is to assess the changes in recorded by the SmartCardia patch (respiratory rate, pulse transit time, heart rate and single ECG trace) during induced ischemia during elective coronary angioplasty procedures.

The secondary objective is to asses whether myocardial ischemia can be predicted and quantified by changes in the parameters recorded by SmartCardia patch (respiratory rate, pulse transit time, heart rate and single ECG trace).

DETAILED DESCRIPTION:
Coronary artery disease and myocardial ischemia are among the leading causes of death and disability in the Westerns countries. Timely and accurate diagnosis of myocardial ischemia at the moment of symptom onset is crucial and often delayed. Portable smart medical devices nowadays offers the possibility of ubiquitous self multi-parametric monitoring. Application of such technologies to timely and autonomous detection of myocardial ischemia could be an effective strategy to an earlier and better treatment of symptomatic coronary artery disease.

The primary objective is to assess the changes in recorded by the SmartCardia patch (respiratory rate, pulse transit time, heart rate and single ECG trace) during induced ischemia during elective coronary angioplasty procedures.

The secondary objective is to asses whether myocardial ischemia can be predicted and quantified by changes in the parameters recorded by SmartCardia patch (respiratory rate, pulse transit time, heart rate and single ECG trace).

SmartWearable devices will be applied 30 minutes before coronary angiography (2/3 devices per-patients would be applied). Percutaneous coronary intervention will be conducted following a given protocol (not influencing patient's treatement):

1. Myocardial ischemia will be measured with the Fractional Flow Reserve (FFR) wire during stent expansion (total artery occlusion caused by balloon inflation). This will have no impact on patients' management as the wire will already have been inserted for the diagnostic procedure and will not have an impact on procedure duration.
2. Recording of a 6 leads electrocardiogram during the ischemia phase, which is anyway always available as part of our routine monitoring system.
3. Patients will systematically be asked for any chest pain or discomfort during ischemia (step which is anyway frequently done in standard procedures), to differentiate between clinical and subclinical ischemia.

At the end of the procedure, the device will be kept during 30 supplementary minutes while the patient is on standard post percutaneous coronary intervention (PCI) surveillance, thus offering measurements during recovery from ischemia.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old patients
* Known coronary artery disease
* Admitted for elective coronary angiography with planned PCI
* Informed consent signed

Exclusion Criteria:

* urgent procedure with possible ongoing ischemia before procedure (i.e. STEMI and NSTEMI in the acute phase)
* Recent acute coronary syndrome (i.e. STEMI and/or NSTEMI <48h or with persistent ST elevation)
* Admission for revascularization of a total chronic occlusion
* Known severe valvular disease
* Decompensated heart-failure
* Decompensated pulmonary condition (such as COPD)
* Pregnant and breast-feeding women
* Patients with prior CABG
* Patients with severe renal failure (eGFR < 30ml/mn)
* Vulnerable patients (minors, participants incapable of judgment or participants under tutelage)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04 (Estimated); Primary Completion 2021-08 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Assessment of Ischemia detection | During Coronary Revascularisation procedure
  Assessment of whether myocardial ischemia induced differences would be recorded by the SmartCardia patch by estimating the effect size observed on each individual parameter recorded by the device for each patient, comparing the values measured on pre- and during-ischemia intervals.

SECONDARY OUTCOMES:
Assessment of ischemia severity | During Coronary Revascularisation procedure
  Establishment of dose-response curve between the recorded parameters by Smart-Cardia and the ischemia severity (based of distal coronary artery pressure)
Model description for coloration between ischemia severity and parameters recorded | During Coronary Revascularisation procedure
  Integration of multiple parameters into a more complex model to increase level of correlation between the recorded parameters and the severity of ischemia

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Switzerland

IPD SHARING:
Plan to Share IPD: No